CLINICAL TRIAL: NCT04460144
Title: Diagnostic Validation Study of a Test Based on the Analysis of the Proteome by Mass Spectrometry for the Diagnosis of Septic Arthritis in Children Under 16 Years of Age.
Brief Title: Rapid Diagnostic Test for Septic Arthritis
Acronym: TDR-Arthrite
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190930; IDRCB 2019-A02427-50 (Other: ANSM)
Record Dates: First submitted 2020-07-01; First posted 2020-07-07 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2021-09

CONDITIONS: Juvenile Idiopathic Arthritis; Arthritis, Septic; Arthritis, Unspecified
MeSH Terms: conditions — Arthritis, Juvenile; Arthritis, Infectious; Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — synovial fluid blood sample stool sample nasal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mass spectrometry — Proteomic analysis

SUMMARY:
Diagnostic Validation Study of a Test Based on the Analysis of the Proteome by Mass Spectrometry for the Diagnosis of Septic Arthritis in Children Under 16 Years of Age

DETAILED DESCRIPTION:
Arthritis is an inflammation of the joints that can have many causes. In children, septic arthritis (SA) is the most common cause of acute arthritis (around 45% of cases). Juvenile Idiopathic Arthritis (JIA) is a disease characterized the presence of arthritis in one or more of unknown origin in children under 16 years of age, lasting more than 6 weeks. It is the most common pediatric rheumatological disease with a prevalence of 16 to 150 cases per 100,000 children. Finally, in approximately 40% of children the origin of acute arthritis remains undetermined (ND arthritis). In this group, all the examinations performed are not in favor of a bacterial origin and the evolution of arthritis do not allow the diagnosis of JIA to be retained and no other disease is found.

During the first few days of arthritis, differentiation between AS and non-septic arthritis is difficult. The available clinical and biological parameters do not allow for easy and rapid differentiation between AS and non-septic arthritis.

This project aims to develop a new diagnostic technique based on molecular analysis of the proteome in the joint puncture fluid.

ELIGIBILITY:
Inclusion Criteria:

* Patients >3 months of age <16 years of age
* Hospitalized for arthritis that started less than 6 weeks ago or patients with diagnosed inflammatory arthritis whose clinical course suggests bacterial superinfection
* Indication of a joint puncture for diagnostic purposes, confirmed by a senior physician after study of all available clinical and biological elements.
* Holders of parental authority who have accepted the participation of their children
* Patients benefiting from a social security scheme (excluding AME)

Exclusion Criteria:

* Contraindications to joint puncture

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with acute arthritis
Sampling Method: Non-Probability Sample
Enrollment: 274 (Actual)
Dates: Start 2021-05-06 (Actual); Primary Completion 2022-10-21 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
Mass spectrometry profile | 15 months
  Proteomics

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich MEINZER, MD-PhD, Principal Investigator — APHP; Stephane BONACORSI, MD-PhD, Study Director — APHP
Locations (1):
- Robert Debre Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided